CLINICAL TRIAL: NCT05454423
Title: Effect of Aquatic Exercise and Traditional Physical Therapy on Gout in Hypertensive Menopausal Women With Hyperuricemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Merit University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A Eon gout
Record Dates: First submitted 2022-06-29; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Intervention Model Description: Aquatic Exercise and traditional physical therapy are effective methods of treatment for gout and hypertension in menopausal women.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aquatic exercise + Traditional physical therapy + anti-hyperuricemia medication (Experimental): consisted of 50 Patients received aquatic exercise and Traditional physical therapy in addition to anti-hyperuricemia medication (a potent purine xanthine oxidase (XO) inhibitor) in therapeutic dose.
  Interventions: Other: the Aquatic exercises +Traditional physical therapy programs +anti-hyperuricemia medication
- traditional physical therapy + anti-hyperuricemia medication (Placebo Comparator): consisted of 50 Patients received traditional physical therapy in addition to anti-hyperuricemia medication (a potent purine xanthine oxidase (XO) inhibitor) in therapeutic dose.
  Interventions: Other: traditional physical therapy + anti-hyperuricemia medication

INTERVENTIONS:
Other: the Aquatic exercises +Traditional physical therapy programs +anti-hyperuricemia medication — -Aquatic exercises: At the beginning of the exercises, aquatic exercises technique was educated to the participants out of water. Then, the aquatic exercises were conducted in a chest warm pool (28-30°C) for 30 minutes, three sessions a week for eight weeks.
  -Traditional physical therapy programs : which included using hot packs (20 minutes), ultrasound (5 minutes), and electrotherapy using TENS (15 minutes) in addition to stretching exercises for the calf, hamstring muscles and big toes and strengthening exercises for the quadriceps muscles for 30 minutes". The stretching exercises were performed in 3 weekly sessions over 8 weeks, each with a 30 second holding and a 30-second relaxation repeated three times. One group of strengthening exercises consisted of 10 repeats with a 5 second holding
  Arms: aquatic exercise + Traditional physical therapy + anti-hyperuricemia medication
Other: traditional physical therapy + anti-hyperuricemia medication — traditional physical therapy programs, which included using hot packs (20 minutes), ultrasound (5 minutes), and electrotherapy using TENS (15 minutes) in addition to stretching exercises for the calf, hamstring muscles and big toes and strengthening exercises for the quadriceps muscles for 30 minutes". The stretching exercises were performed in 3 weekly sessions over 8 weeks, each with a 30 second holding and a 30 second relaxation repeated three times. One group of strengthening exercises consisted of 10 repeats with a 5 second holding17.
  Arms: traditional physical therapy + anti-hyperuricemia medication

SUMMARY:
Aquatic Exercise and traditional physical therapy are effective methods of treatment for gout and hypertension in menopausal women.

DETAILED DESCRIPTION:
Menopause is defined as a point in time 12 months after a woman's last period. During the menopausal transition, changes in estrogen and progesterone levels affect not only vasomotor symptoms, sexual dysfunction, osteoporosis, and cardiovascular disease (CVD), but also uric acid level1. An association between menopausal status and hyperuricemia has been previously examined. A study using the Third National Health and Nutrition Examination Survey showed a positive and independent association of menopause with hyperuricemia and gout. It's believed that estrogen has a protective effect that is removed at menopause, thus accounting for the rise in gout in women who are postmenopausal2.

Hyperuricemia is a common biochemical abnormality resulting from excessive uric acid production or impaired clearance of uric acid. Although its pathophysiology is not fully understood, genetic, comorbid disease-related, and environmental (drug, diet, and toxic exposure-induced) factors are involved in hyperuricemia3.

Gout is a multifactorial disease caused by hyperuricemia and monosodium urate crystals deposition. Pain typically comes on rapidly, reaching maximal intensity in less than 12 hours. The joint at the base of the big toe is affected in about half of cases4.

ELIGIBILITY:
Inclusion Criteria:

* 100 patients with gout

  * Age between 45 -65 years
  * Cooperative patient.
  * A physician referred all patients with the diagnosis of gout

Exclusion Criteria:

* history of kidney disease such as chronic kidney disease, Cancer patients. Smokers Patients with chronic heart disease.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Serum uric acid level before and after treatment for both groups (A and B): Table 2: Mean values for Serum uric acid level before and after treatment for both groups (A and B). | 2 week before and 2 week after
  a sample of blood was used to assess the level of uric acid in the blood for both groups A & B before and after treatment
Visual analogue scale before and after treatment for both groups (A and B): Chicago, Illinois, USA). The P-value is the degree of significance. A P value less than or equal to 0.05 was considered to be significant. | 2 week before and 2 week after
  consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be. The patient was asked to mark her pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain intensity .
The Borg Rating of Perceived Exertion (RPE) scale | 2 week before and 2 week after
  will be used to measure the level of exertional effort for both groups A & B before and after treatment
Digital blood pressure monitor | 2 week before and 2 week after
  It measures blood pressure (systolic & diastolic) quickly, is easy to use, reliable, and convenient to carry. The monitor has a display that shows systolic blood pressure and diastolic blood pressure. The machine comes with an arm cuff with an air tube and an air jack for connecting the cuff to the machine

REFERENCES:
- [Background] Derby CA, Crawford SL, Pasternak RC, Sowers M, Sternfeld B, Matthews KA. Lipid changes during the menopause transition in relation to age and weight: the Study of Women's Health Across the Nation. Am J Epidemiol. 2009 Jun 1;169(11):1352-61. doi: 10.1093/aje/kwp043. Epub 2009 Apr 8. PMID 19357323
- [Background] Richette P, Bardin T. Gout. Lancet. 2010 Jan 23;375(9711):318-28. doi: 10.1016/S0140-6736(09)60883-7. Epub 2009 Aug 17. PMID 19692116
- [Background] Dalbeth N, Merriman TR, Stamp LK. Gout. Lancet. 2016 Oct 22;388(10055):2039-2052. doi: 10.1016/S0140-6736(16)00346-9. Epub 2016 Apr 21. PMID 27112094